CLINICAL TRIAL: NCT05937906
Title: Phase Ib/II Clinical Trial Evaluating the Safety and Efficacy of Chemoimmunotherapy Plus Short Course of Mek Inhibitor in First Line of Treatment of Metastatic Non Squamous Non Small Cell Lung Adenocarcinoma With PDL1 < 50 %.
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of Chemoimmunotherapy Plus Short Course of Mek Inhibitor in First Line of Treatment of Metastatic Non Squamous Non Small Cell Lung Adenocarcinoma With PDL1 < 50 %.
Acronym: IMMUNOMEK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508477-87-00
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: locally advanced or metastatic; non squamous non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Phase 1 (escalation dose)
  * Level 1: mirdametinib 4 mg twice/day for 7 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab until progression (3-6 patients)
  * Level 2: mirdametinib 4 mg twice/day for 14 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab until progression (3-6 patients)
  * Level 3: mirdametinib 6 mg twice/day for 7 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab until progression (3-6 patients)
  * Level 4: mirdametinib 6 mg twice/day for 14 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab until progression (3-6 patients)
  Phase 2 (randomized)
  * Standard arm : Carboplatin/pemetrexed/pembrolizumab for the first 4 cycles until progression (26 patients)
  * Experimental arm : Carboplatin/pemetrexed/pembrolizumab + mirdametinib for the first 4 cycles until progression (52 patients)
Masking Description: Non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase I - Level 1 (Experimental): Mirdametinib 4 mg twice/day for 7 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab.
  Pemetrexed/pembrolizumab until progression Number of participants : 3 to 6 patients
  Interventions: Drug: Phase I - Mirdametinib - Level 1
- Phase I - Level 2 (Experimental): Mirdametinib 4 mg twice/day for 14 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab.
  Pemetrexed/pembrolizumab until progression Number of participants : 3 to 6 patients
  Interventions: Drug: Phase I - Mirdametinib - Level 2
- Phase I - Level 3 (Experimental): Mirdametinib 6 mg twice/day for 7 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab.
  Pemetrexed/pembrolizumab until progression Number of participants : 3 to 6 patients
  Interventions: Drug: Phase I - Mirdametinib - Level 3
- Phase I - Level 4 (Experimental): Mirdametinib 6 mg twice/day for 14 days per cycle for the 4 first cycles + carboplatin/pemetrexed/pembrolizumab.
  Pemetrexed/pembrolizumab until progression Number of participants : 3 to 6 patients
  Interventions: Drug: Phase I - Mirdametinib - Level 4
- Phase II - Standard arm (No Intervention): Carboplatin / Pemetrexed / Pembrolizumab for the first 4 cycles
- Phase II - Experimental arm (Experimental): Carboplatin / Pemetrexed / Pembrolizumab + mirdametinib for the first 4 cycles
  Interventions: Drug: Phase II - Mirdametinib

INTERVENTIONS:
Drug: Phase I - Mirdametinib - Level 1 — Mirdametinib 4 mg twice/day for 7 days per cycle
  Arms: Phase I - Level 1
Drug: Phase II - Mirdametinib — For phase 2 : Randomisation with 2 arm : Standard arm and experimental arm
  Arms: Phase II - Experimental arm
Drug: Phase I - Mirdametinib - Level 2 — Mirdametinib 4 mg twice/day for 14 days per cycle
  Arms: Phase I - Level 2
Drug: Phase I - Mirdametinib - Level 3 — Mirdametinib 6 mg twice/day for 7 days per cycle
  Arms: Phase I - Level 3
Drug: Phase I - Mirdametinib - Level 4 — Mirdametinib 6 mg twice/day for 14 days per cycle
  Arms: Phase I - Level 4

SUMMARY:
Monocentric study composed by 2 steps :

1. First step is a phase I with the aim of establish the recommended dose of mirdametinib administration (2 or 4 mg twice a day for 7 or 14 days per cycle for the 4 first of carboplatin/pemetrexed/pembrolizumab treatment)
2. Second step is a non comparative randomized (2:1) phase II trial testing the recommended dose of mirdametinib administration. The aim is the efficacy and safety of short course of mirdametinib treatment for the 4 first cycles of the carboplatin/pemetrexed/pembrolizumab treatment.

DETAILED DESCRIPTION:
1) Phase I (15-24 patients) Using a classical "3+3 design": The phase I will included a maximum 24 patients. 3 patients will be included in dose level 1, if not DLT occurs 3 patients will be included in level 2. If 1 DLT occurs 3 additional patients will be included; if 2 or more DLT occurs the trial will be stopped. At level 2 if no DLT occurs RP2D 3 patients will be included at level 3; If 1 DLT occurs 3 additional patients will be included; if 2 or more DLT occurs RP2D will be level 1. Similar rules will be applied for level 3 and 4. In absence of DLT CXCL10 and PD-L1, CD8 immune infiltrates and immunoscore IC (CD8-PDL1 dual markers) at baseline and 6 weeks, and clinical efficacy will be presented to IDMC for definition of RP2D. At the end of phase I inclusion toxicity, efficacy data and biological data (CXCL10 seric and IHC expression and PD-L1, CD8 immune infiltrates and immunoscore IC (CD8-PDL1 dual markers) at baseline and 6 weeks, PK and PK/PD data will be presented to IDMC to validate RP2D.

* 3 +/- 3 patients for level 1 (mirdametinib 4 mg twice/ 7 days)
* 3 +/- 3 patients for level 2 (mirdametinib 4 mg twice/ 14 days)
* 3 +/- 3 patients for level 3 (mirdametinib 6 mg twice/ 7 days)
* 3 +/- 3 patients for level 4 (mirdametinib 6 mg twice/ 14 days)

PHASE II (78 patients) Sample size calculation was performed using PASS v13. In keynote 189 response rate in PD-L1 <50% was 40% (28). A 3-month overall response rate (ORR) of 40% is considered unacceptable (P0=40%). The study team expect an ORR of 55% in the experiment arm (P1=55%, acceptable ORR).

Using a single stage design (A Hern, exact test) with unilateral α=10%, power=80%, 50 patients are needed for the primary endpoint analysis in the experimental arm. With 5% of non-evaluable patients, 52 patients will be included in this arm. With a 2:1 randomization the control arm will include 26 patients. A total of 78 subjects are then needed in the phase 2 part.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
* Patients must be diagnosed with a metastatic or locally advanced non squamous non-small cell lung cancer
* Absence of previous treatment for or locally advanced or metastatic non-small cell lung cancer. Previous adjuvant therapy is allowed if > 12 months from the last injection
* Age >18 years at time of study entry
* Performance status ECOG of 0 or 1
* Life expectancy ≥ 6 months
* PD-L1<50% using TPS scoring
* At least one lesion measurable as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1) that can be accurately assessed at baseline and is suitable for repeated assessment
* Body weight >30 kg
* Adequate normal organ and marrow function as defined below:
* Adequate cardiac function:

(QTc < 450 msec on baseline ECG, using the Fridericia correction cQTcF formula) or other clinically significant ventricular or atrial arrhythmia.

Left ventricular ejection fraction (LVEF) ≥ 50%

* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patient affiliated to a social security regimen or beneficiary of the same according
* Validation of the quality and quantity of the tumoral material at inclusion (existing material dated less than one month and/or fresh biopsy).
* Patient is willing to perform the fresh biopsies mandatory for the protocol:

Phase I: A mandatory fresh biopsy of 4 samples at inclusion and after Cycle 2 (betweenC2J7 and C2J14) Phase II: A mandatory fresh biopsy. of 4 samples at inclusion. Second biopsy at 4-5 weeks after treatment initiation is optional.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 2 months
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Presence of EGFR, ROS or ALK targetable mutations
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, ototoxicity, vitiligo, and the laboratory values defined in the inclusion criteria. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable before the first dose of study drug
* Major surgical procedure within 28 days prior to therapy initiation IP. Note: Local surgery of isolated lesions for palliative intent is acceptable. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48 hour interval must be maintained before the first dose of study drug
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea or malabsorption syndrome).
* History of allogenic organ, bone marrow or double umbilical cord blood transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

Patients with vitiligo or alopecia Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active disease in the last 5 years may be included but only after consultation with the study physician Patients with celiac disease controlled by diet alone

* History of glaucoma, any retinal pathology considered to be a risk factor for central serous retinopathy, retinal vein occlusion (RVO) or neovascular macular degeneration. Also, any risk factors for RVO as intraocular pressure (IOP) >21, uncontrolled blood glucose
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease. Any uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (including history of myocardial infarction within 3 months, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, or any cardiac arrhythmias, e.g, ventricular, supraventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening) uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high Resolution Computed Tomography (HRCT) sacan or any psychiatric disorder that prohibits obtaining informed consent.
* Currently taking medications with known risk of prolonging the QT interval or inducing Torsades de Pointes
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, cQTcF prolongation >450ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML
* History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Patient with symptomatic central nervous system (CNS) metastases
* History of active primary immunodeficiency or Immunocompromised patients e.g, patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of immunotherapy. The following are exceptions to this criterion:

Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

* Receipt of live or live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine (yellow fever vaccination is forbidden) whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of treatment. (Contraceptive requirements: Male patients must use a condom during treatment and for 3 months after the last dose when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.)
* Known allergy or hypersensitivity to any of the study drugs or any of the study drugs excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Safety will be evaluated using Dose Limiting Toxicities (DLT) | Until progression, an average of 10 months
  DLT is defined as any of the following toxicities occurring during the first 21 days after administration of the first dose. Adverse events (AEs) will be defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges-François Leclerc, Dijon, Burgundy, France